CLINICAL TRIAL: NCT01426347
Title: Vitamin Therapy in Rheumatoid Arthritis
Brief Title: Treatment of Vitamin D Deficiency in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VDRA
Record Dates: First submitted 2011-08-29; First posted 2011-08-31 (Estimated); Results first posted 2017-03-20 (Actual); Last update posted 2017-03-20 (Actual); Status verified 2017-01

CONDITIONS: Rheumatoid Arthritis; Vitamin D Deficiency
Keywords: Rheumatoid Arthritis; Vitamin D deficiency; Disability
MeSH Terms: conditions — Arthritis, Rheumatoid; Vitamin D Deficiency | interventions — Ergocalciferols; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo group (Placebo Comparator): RA Patients with vitamin D deficiency will be randomized to placebo and active intervention arms.
  Patients in the placebo arm will receive I placebo pill per week for 16 weeks. After completing this arm, they will cross-over to the active treatment arm.
  Interventions: Drug: Placebo sugar pill; Drug: Ergocalciferol
- Ergocalciferol (Active Comparator): Patients with vitamin D deficiency will be randomized to either active or placebo group. In the active group, patients will receive ergocalciferol 50,000 IU per week for 16 weeks.
  Interventions: Drug: Ergocalciferol

INTERVENTIONS:
Drug: Placebo sugar pill — Intervention includes 1 sugar pill once a week for 16 weeks dispensed as a capsule.
  Other Names: Placebo
  Arms: placebo group
Drug: Ergocalciferol — Ergocalciferol 50,000 IU per week for 16 weeks
  Other Names: Vitamin D

SUMMARY:
The purpose of this study is to investigate the effect of vitamin D repletion on disease activity and disability in patients with rheumatoid arthritis.

The investigators hypothesize that rheumatoid arthritis (RA) patients with vitamin D deficiency have greater disease activity and disability, compared to RA patients with normal vitamin D levels. The investigators also hypothesize that vitamin D treatment in these deficient patients will result in a decrease in RA disease activity and disability.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid Arthritis diagnosed according to American College of Rheumatology (ACR) criteria
* ages 18-75 years

Exclusion Criteria:

* Diagnosis of any other autoimmune disease:

such as Lupus, Scleroderma, Myositis, Sjogren's Syndrome, Vasculitis'

* Having any of the following conditions with in the last 6 months Hypercalcemia, Hyperparathyroidism, Active tuberculosis (TB), Lymphoma or any other type of cancer, Sarcoidosis, Seizure, Stroke
* Severe heart problems
* Kidney failure requiring dialysis treatment
* Liver failure or cirrhosis of the liver
* Poorly controlled hypertension
* current uncontrolled Depression, Bipolar Disorder, or other Psychiatric illness
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2009-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Uzma J Haque, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One hundred thirty-nine (139) participants were enrolled for visit 1, and blood was drawn to determine vitamin D levels. Eighty-three (83) were vitamin D deficient by criteria, vitamin D < 30 nanogram/milliliter (ng/ml), and entered the randomized controlled trial. The remaining 56 exited the study because they were vitamin D sufficient.
Groups:
- Placebo Group: Rheumatoid Arthritis (RA) patients with vitamin D deficiency will be randomized to placebo and active intervention arms.
  Patients in the placebo arm will receive I placebo pill per week for 16 weeks. After completing this arm, they will cross-over to the active treatment arm.
  Placebo sugar pill: Intervention includes 1 sugar pill once a week for 16 weeks dispensed as a capsule.
Period: Overall Study
Arm/Group | Placebo Group | Ergocalciferol
Started | 41 | 42
Completed | 34 | 39
Not Completed | 7 | 3
Not completed — Lost to Follow-up | 0 | 3
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo Group: RA Patients with vitamin D deficiency will be randomized to placebo and active intervention arms.
  Patients in the placebo arm will receive I placebo pill per week for 16 weeks. After completing this arm, they will cross-over to the active treatment arm.
  Placebo sugar pill: Intervention includes 1 sugar pill once a week for 16 weeks dispensed as a capsule.
- Total: Total of all reporting groups
Arm/Group | Placebo Group | Ergocalciferol | Total
Number analyzed (Participants) | 41 | 42 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (13.5) | 52.2 (12.2) | 52.5 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 36 | 69
  Male | 8 | 6 | 14
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 32 | 31 | 63
  Non-caucasian | 9 | 11 | 20

OUTCOME MEASURES:

1. Primary Outcome: Disease Activity Score (DAS) 28
Description: We measured disease activity as measured by DAS 28 at baseline and at the completion of Randomized Controlled trial, both in the placebo and the active treatment group.
  We used DAS-28 scores to indicate disease activity. The DAS -28 scale has a minimum of 0 and a maximum of 10, with higher numbers indicating higher disease activity.
  We used the following cut-offs: Remission (< 2.6), low disease activity (< 3.2), moderate disease activity (< 5.1) and high disease activity (> 5.1).
Time Frame: Baseline and 16 weeks (end of Randomized Controlled Trial (RCT))
Measure: Mean (Standard Deviation); unit: composite score
Arm/Group | Placebo Group | Ergocalciferol
Number analyzed (Participants) | 41 | 42
composite score
  Baseline | 3.4 (1.5) | 2.8 (1.3)
  16 weeks (end of RCT) | 3.5 (1.5) | 3.1 (1.3)

2. Secondary Outcome: Physical Function as Measured by Arthritis Impact Measurement Scales - Short Form (AIMS2 - SF)
Description: In each dimension and component of AIMS2-SF, item scores are from 0 to 10 with 10 being worst health.
Time Frame: Baseline and 16 weeks (end of RCT)
Population: For placebo, analysis is based on 26 at baseline and 33 at the end of RCT For treatment, analysis is based on 27 at baseline and 38 at the end of RCT
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Group | Ergocalciferol
Number analyzed (Participants) | 33 | 38
units on a scale
  Baseline | 1.9 (1.3) | 1.7 (1.6)
  16 weeks (end of RCT) | 1.9 (1.5) | 1.6 (2.1)

ADVERSE EVENTS:
Arm/Group | Placebo Group | Ergocalciferol
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/42
Other Adverse Events (participants affected / at risk) | 0/41 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes